CLINICAL TRIAL: NCT00734331
Title: Micro Ribonucleic Acid (RNA) as Cholinergic Tone and Inflammatory Regulator in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, michal roll, MicroRNA-132 Modulates Cholinergic Signaling and Inflammation in Human Inflammatory Bowel Disease, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-NM-300-CTIL
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; micro RNA; cholinergic tone; inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, colonic tissue, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBD: Inflammatory bowel disease patients
- Control: Average risk patients undergoing screening colonoscopy

SUMMARY:
There is a reciprocal relationship between the central nervous system and the immune system. Stimulation of the vagus nerve results in secretion of acetylcholine (Ach) which decreases secretion of pro-inflammatory cytokines. Acetylcholine esterase is an enzyme that neutralizes Ach and thus, involves in regulation of Ach levels, and in the cholinergic tone and inflammatory state.

MicroRNAs (miRs) are evolutionarily conserved, RNAs that regulate gene expression. The investigators hypothesized that miRs controlling systemic communication processes function in one tissue in response to signals (i.e. neuronal, hormonal or others) from another.

Specifically, the investigators hypothesized that miRs control the inflammatory response in inflammatory bowel diseases through regulation of expression of messenger RNA of AchE.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease patients under going colonoscopy

Exclusion Criteria:

* Debilitated patients who need an apotropsy
* Age < 18 or age > 75
* Pregnant women
* Evidence of previous or current cancer
* Inflammatory disease other than IBD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients- inflammatory bowel disease patients under going colonoscopy controls- average risk patients without inflammation under going colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Elevated expression of specific micro RNAs that regulate the expression of the enzyme Acetylcholine esterase in inflammatory bowel disease patients compared to healthy controls. | one year

SECONDARY OUTCOMES:
A statistically significant relation between micro RNA expression and disease activity and inflammatory indices | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel